CLINICAL TRIAL: NCT05791773
Title: Robotic Total Knee Arthroplasty Anesthesia Management: Retrospective Study
Brief Title: Robotic Total Knee Arthroplasty Anesthesia Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Umut Kara, Associate Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2022-98
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis; Joint Diseases; Anesthesia
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group rTKA (robotic total knee arthroplasty): the robot assisted total knee arthroplasty
  Interventions: Procedure: the robot assisted total knee arthroplasty
- Group cTKA (conventional total knee arthroplasty): the conventional jig-based total knee arthroplasty
  Interventions: Procedure: the conventional jig-based total knee arthroplasty

INTERVENTIONS:
Procedure: the robot assisted total knee arthroplasty — the robot assisted total knee arthroplasty
  Groups: Group rTKA (robotic total knee arthroplasty)
Procedure: the conventional jig-based total knee arthroplasty — the conventional jig-based total knee arthroplasty
  Groups: Group cTKA (conventional total knee arthroplasty)

SUMMARY:
Robotic arthroplasty is increasing in acceptance on a global scale as a result of advancements in orthopedic surgery technology.

The investigators aimed to share our anesthesia management experience as well as compare robotic unilateral total knee arthroplasty with conventional surgical technique in this retrospective study.

DETAILED DESCRIPTION:
This study was approved by the ethics committee of a tertiary academic hospital.

The following criteria were used to assess inclusion: ASA physical status I-III patients aged 40-85 years, elective unilateral total knee arthroplasty (TKAs) performed by a single senior orthopedic surgeon and orthopedic team under combined spinal epidural anesthesia (CSEA) between January 2021 and January 2023. Exclusion criteria included urgent surgery, bilateral surgery, previous surgery, missing data, and being lost to follow-up during the perioperative period. Data was collected from the hospital's electronic database records, patient files, and anesthesia charts.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Between 40-85 years
* Elective unilateral TKAs which were performed by a single senior orthopedic surgeon
* Between January 2021 and January 2023 under CSEA.

Exclusion Criteria:

* Urgent surgery
* Bilateral surgery
* Previous surgery
* Missing data and lost to follow-up in the perioperative period

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with American Society of Anesthesiologists (ASA) physical status I-III and elective unilateral TKAs between the ages of 40 and 85 will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Time | Only in surgery time, an average of 3 hours
  The duration of surgical procedures

SECONDARY OUTCOMES:
Complications | After the end of surgery, in the first 1-month follow-up
  Perioperative complications rates
Hospital discharge time | Time from discharge from PACU to discharge from hospital, an average of 96 hours
  Time from the beginning of the operation to the discharge of hospital

IPD SHARING:
Plan to Share IPD: Undecided